CLINICAL TRIAL: NCT02546674
Title: A Phase IV Single Arm, Multicenter, Open-label Study Assessing Deep Molecular Response in Adult Patients With Newly Diagnosed Philadelphia Chromosome Positive CML in Chronic Phase After Two Years of Treatment With Nilotinib 300mg BID
Brief Title: Study Assessing Deep Molecular Response in Adult Patients With CML in Chronic Phase Treated With Nilotinib Firstline.
Acronym: NILOdeepR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAMN107ADE20; 2015-000968-34 (EudraCT Number)
Record Dates: First submitted 2015-09-09; First posted 2015-09-11 (Estimated); Results first posted 2022-07-22 (Actual); Last update posted 2022-07-22 (Actual); Status verified 2022-03

CONDITIONS: Chronic Myeloid Leukemia
Keywords: Chronic Myeloid Leukemia; Nilotinib; Molecular Response; MR4.5
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — nilotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nilotinib (Experimental): Participants with newly diagnosed CML in chronic phase received nilotinib 300 mg BID for 24 months
  Interventions: Drug: Nilotinib

INTERVENTIONS:
Drug: Nilotinib — A daily dose of 300 mg was given to all participants as two 150 mg capsules BID. The prescription of study drug was not study dependent and followed medical needs of the participant only. The study treatment was administered for 24 months.
  Other Names: AMN107

SUMMARY:
The main purpose of this study was to evaluate the rate of deep molecular response (MR4.5) after 24 months of therapy with nilotinib in newly diagnosed patients with chronic phase chronic myeloid leukemia (CML) using EUTOS (European Treatment and Outcome Study for CML)-standardized laboratories. All participants received nilotinib 300 mg twice daily (BID).

DETAILED DESCRIPTION:
This was a Phase IV open-label, multi-center, single-arm study in participants with newly diagnosed Philadelphia chromosome positive (Ph+) CML in chronic phase for who nilotinib is the appropriate treatment at the discretion of the investigator.

A screening period of 2 weeks was used to assess eligibility and to taper participants off disallowed medications. Participants whose eligibility was confirmed entered a 24 months treatment phase with nilotinib 300mg BID. Nilotinib was prescribed by the investigator according to the individual needs of the participants.

ELIGIBILITY:
Key Inclusion Criteria:

* Patients with newly diagnosed (within 6 months) Philadelphia chromosome positive CML in chronic phase
* Patients must be previously untreated for CML with the exception of 6 months treatment with hydroxyurea and a maximum of 6 weeks treatment with imatinib
* Adequate end organ function
* Normal serum levels ≥ lower limit of normal (LLN) of potassium, magnesium, total calcium corrected for serum albumin or phosphorus, or correctable to within normal limits with supplements, prior to the first dose of study medication.

Key Exclusion Criteria:

* Known impaired cardiac function like long QT syndrome, history of myocardial infarction or unstable angina in the past 12 months.
* Patients who are pregnant or breast feeding.

Other inclusion/exclusion criteria might apply

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 171 (Actual)
Dates: Start 2016-02-18 (Actual); Primary Completion 2021-02-23 (Actual); Study Completion 2021-03-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (61):
- Germany (61):
  - Novartis Investigative Site, Mannheim, Baden-Wurttemberg
  - Novartis Investigative Site, Herne, North Rhine-Westphalia
  - Novartis Investigative Site, Lübeck, Schleswig-Holstein
  - Novartis Investigative Site, Aschaffenburg
  - Novartis Investigative Site, Augsburg
  - Novartis Investigative Site, Bad Mergentheim
  - Novartis Investigative Site, Bad Reichenhall
  - Novartis Investigative Site, Bad Saarow
  - Novartis Investigative Site, Bad Soden
  - Novartis Investigative Site, Bamberg
  - Novartis Investigative Site, Bayreuth
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Biberach
  - Novartis Investigative Site, Bremerhaven
  - Novartis Investigative Site, Chemnitz
  - Novartis Investigative Site, Cologne
  - Novartis Investigative Site, Donauwörth
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Düsseldorf
  - Novartis Investigative Site, Erfurt
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Georgsmarienhütte
  - Novartis Investigative Site, Giessen
  - Novartis Investigative Site, Goslar
  - Novartis Investigative Site, Göppingen
  - Novartis Investigative Site, Halberstadt
  - Novartis Investigative Site, Halle
  - Novartis Investigative Site, Halle S
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Heidelberg
  - Novartis Investigative Site, Jena
  - Novartis Investigative Site, Kassel
  - Novartis Investigative Site, Kiel
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Magdeburg
  - Novartis Investigative Site, Memmingen
  - Novartis Investigative Site, Minden
  - Novartis Investigative Site, Moers
  - Novartis Investigative Site, Mutlangen
  - Novartis Investigative Site, Mülheim
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Münster
  - Novartis Investigative Site, Nuremberg
  - Novartis Investigative Site, Oldenburg
  - Novartis Investigative Site, Paderborn
  - Novartis Investigative Site, Passau
  - Novartis Investigative Site, Potsdam
  - Novartis Investigative Site, Rostock
  - Novartis Investigative Site, Rotenburg (Wümme)
  - Novartis Investigative Site, Saarbrücken
  - Novartis Investigative Site, Schorndorf
  - Novartis Investigative Site, Schwäbisch Hall
  - Novartis Investigative Site, Schweinfurt
  - Novartis Investigative Site, Tübingen
  - Novartis Investigative Site, Velbert
  - Novartis Investigative Site, Westerstede
  - Novartis Investigative Site, Wiesbaden
  - Novartis Investigative Site, Wilhelmshaven
  - Novartis Investigative Site, Wolfsburg
  - Novartis Investigative Site, Worms
  - Novartis Investigative Site, Würzburg

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- See also: Related Info — http://www.leukaemie-online.de/studien/70-studie-erstlinie/1198-nilo-deep-r-studie

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted across 73 centers in 1 country (Germany).
Pre-assignment Details: A total of 179 participants were screened in this study of which 8 discontinued screening phase and 171 participants were enrolled in the study
Groups:
- Nilotinib: Participants with newly diagnosed CML in chronic phase received nilotinib 300 mg BID
Period: Overall Study
Arm/Group | Nilotinib
Started | 171
Completed | 123
Not Completed | 48
Not completed — Adverse Event | 19
Not completed — Death | 1
Not completed — Lost to Follow-up | 1
Not completed — Physician Decision | 13
Not completed — Pregnancy | 1
Not completed — Progressive Disease | 2
Not completed — Protocol Deviation | 2
Not completed — Subject/Guardian Decision | 6
Not completed — Withdrawal of Informed Consent | 3

BASELINE CHARACTERISTICS:
Arm/Group | Nilotinib
Number analyzed (Participants) | 171
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55.2 (13.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 63
  Male | 108
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 170
  Asian | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Deep Molecular Response MR4.5 at 24 Months of Study Treatment
Description: Percentage of participants who were in deep molecular response MR4.5 (IS) at 24 months measured in a standardized EUTOS (European Treatment and Outcome Study for CML) MR4.5 laboratory. MR4.5 was defined as either (i) detectable disease ≤ 0.0032% BCR-ABL (fusion gene from breakpoint cluster region and Abelson genes) (IS) or (ii) undetectable disease in cDNA with 32000-99999 ABL1 transcripts or 77000-239999 glucuronidase beta (GUSB) transcripts.
  Responders: Participants with a MR4.5 at 24 months, or if the assessment at this time point was missing, with a MR4.5 at 21 months Non-responders: Participants dropping out early or not providing sufficient data for any other reason. Participants who achieved MR4.5 before 24 months, but was no longer in MR4.5 at 24 months or progressed (or was no longer in MR4.5 at 21 months if evaluation at 24 months was missing).
  Confidence intervals were calculated based on the Exact Clopper-Pearson method.
Time Frame: Month 24 and Month 21 (if assessment at Month 24 was missing)
Population: Full Analysis Set (FAS): all participants who entered study and received at least one dose of study drug and had at least one post-baseline assessment of the primary efficacy variable. Only participants in the FAS with typical BCR-ABL transcripts (b2a2 and/or b3a2) were included in the analysis. Participants with atypical transcripts were excluded from the analysis, because their transcripts could not be used for molecular response determination
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Nilotinib
Number analyzed (Participants) | 156
Percentage of participants | 35.3 [27.79 to 43.30]

2. Secondary Outcome: Percentage of Participants With MR4 at 24 Months of Study Treatment.
Description: Percentage of participants with MR4 at 24 months of study treatment. MR4 (IS) is defined as either (i) detectable disease ≤0.01% BCR-ABL by IS or (ii) undetectable disease in cDNA with 10000 - 31999 ABL1 transcripts or 24000 - 76999 GUSB transcripts.
  Confidence intervals were calculated based on the Exact Clopper-Pearson method.
Time Frame: Month 24
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Nilotinib
Number analyzed (Participants) | 156
Percentage of participants | 44.9 [36.91 to 53.03]

3. Secondary Outcome: Percentage of Participants With Major Molecular Response (MMR) at 12 Months of Study Treatment
Description: Percentage of participants with MMR at 12 months of study treatment. MMR is defined as ≤ 0.1% BCR-ABL by IS, or equivalent to ≥ 3 log reduction of BCR-ABL transcript from standardized baseline.
  Confidence intervals were calculated based on the Exact Clopper-Pearson method.
Time Frame: Month 12
Population: FAS: all participants who entered study and received at least one dose of study drug and had at least one post-baseline assessment of the primary efficacy variable. Only participants in the FAS with typical BCR-ABL transcripts (b2a2 and/or b3a2) were included in the analysis. Participants with atypical transcripts were excluded from the analysis, because their transcripts could not be used for molecular response determination
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Nilotinib
Number analyzed (Participants) | 156
Percentage of participants | 60.3 [52.12 to 67.99]

4. Secondary Outcome: Percentage of Participants With Complete Cytogenetic Response (CCyR) at 6 Months of Study Treatment
Description: Percentage of participants with CCyR at 6 months of study treatment. Cytogenetic response was assessed as the percentage of Philadelphia positive (Ph+) metaphases in the bone marrow (a review of a minimum of 20 metaphases was required). CCyR was defined as a value of 0% Ph+ metaphases in bone marrow.
  Confidence intervals were calculated based on the Exact Clopper-Pearson method.
Time Frame: Month 6
Population: FAS: all participants who entered study and received at least one dose of study drug and had at least one post-baseline assessment of the primary efficacy variable. Only participants with review of a minimum of 20 metaphases at month 6 were included in the analysis
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Nilotinib
Number analyzed (Participants) | 19
Percentage of participants | 89.5 [66.86 to 98.70]

5. Secondary Outcome: Progression-free Survival
Description: Progression-free survival is defined as the time from the date of start of study treatment to the date of the first documented disease progression to accelerated phase (AP)/ blast crisis (BC) or death from any cause, whichever is earlier.
  AP is defined as:
  * 15% blasts in the peripheral blood or one marrow aspirate, but <30% blasts in both the peripheral blood and bone marrow aspirate
  * 30% blasts plus promyelocytes in peripheral blood or bone marrow aspirate
  * 20% basophils in the peripheral blood or bone marrow Thrombocytopenia (<100 x 109/Liter) that is unrelated to therapy Evidence of clonal evolution
  BC is defined as:
  ≥ 30% blasts in peripheral blood or bone marrow aspirate Appearance of extramedullary involvement other than hepatosplenomegaly proven by biopsy (i.e., chloroma)
Time Frame: From date of start of treatment to first documented disease progression to AP/ BC or death, assessed up to 24 months
Population: FAS: all participants who entered study and received at least one dose of study drug and had at least one post-baseline assessment of the primary efficacy variable.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Nilotinib
Number analyzed (Participants) | 162
Months | NA [NA to NA] — NA: Not estimable due to the very low number of events reported

6. Secondary Outcome: Time to Progression to AP/BC
Description: Time to progression to AP/BC is defined as the time from the date of start of study treatment to the date of earliest transformation to AP/BC, or CML-related death.
  AP is defined as:
  * 15% blasts in the peripheral blood or one marrow aspirate, but <30% blasts in both the peripheral blood and bone marrow aspirate
  * 30% blasts plus promyelocytes in peripheral blood or bone marrow aspirate
  * 20% basophils in the peripheral blood or bone marrow Thrombocytopenia (<100 x 109/L) that is unrelated to therapy Evidence of clonal evolution (with consensus of SC only)
  BC is defined as:
  ≥ 30% blasts in peripheral blood or bone marrow aspirate Appearance of extramedullary involvement other than hepatosplenomegaly proven by biopsy (i.e., chloroma)
Time Frame: From the date of start of study treatment to the date of earliest transformation to AP/BC or CML-related death, assessed up to 24 months
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Nilotinib
Number analyzed (Participants) | 162
Months | NA [NA to NA] — NA: Not estimable due to the very low number of events reported

7. Secondary Outcome: Change From Baseline in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core-30 (EORTC QLQ-C30): Global Health Status (GHS)/Quality of Life (QoL)
Description: The EORTC QLQ-C30 is a patient completed 30 item questionnaire that is composed of both multi-item scales and single-item measures. These include five functional scales, three symptom scales, six single items and a GHS/QoL scale.
  The GHS/QoL scale has 7 possible scores of responses (1=very poor to 7=excellent). Scores were averaged and transformed to 0 to 100. Higher scores indicate better quality of life.
  A positive change from Baseline indicates improvement.
Time Frame: Baseline, month 3, month 6, month 12, month 18 and month 24
Population: FAS: all participants who entered study and received at least one dose of study drug and had at least one post-baseline assessment of the primary efficacy variable. Number analyzed indicated number of participants with available data for this outcome measure at specified timepoints.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Nilotinib
Number analyzed (Participants) | 162
Score on a scale
  Month 3: number analyzed (Participants) | 113
  Month 3 | 5.1 (22.39)
  Month 6: number analyzed (Participants) | 109
  Month 6 | 6.3 (20.29)
  Month 12: number analyzed (Participants) | 99
  Month 12 | 6.0 (25.09)
  Month 18: number analyzed (Participants) | 85
  Month 18 | 4.0 (26.34)
  Month 24: number analyzed (Participants) | 38
  Month 24 | 2.4 (27.05)

8. Secondary Outcome: Change From Baseline in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core-30 (EORTC QLQ-C30): Physical Functioning
Description: The EORTC QLQ-C30 is a patient completed 30 item questionnaire that is composed of both multi-item scales and single-item measures. These include five functional scales, three symptom scales, six single items and a global health status/QoL scale.
  For the physical functioning scale, participants self-rated levels of difficulty in doing strenuous activities, taking a walk, how much they needed to stay in bed or a chair, or needed help with eating, dressing, bathing, using the toilet. The physical functioning scale had 4 possible scores (1=not at all, 2=a little, 3=quite a bit, 4=very much). Scores were averaged and transformed to 0 to 100. Higher scores indicate better functioning. A positive change from baseline indicates improvement in physical functioning.
Time Frame: Baseline, month 3, month 6, month 12, month 18 and month 24
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Nilotinib
Number analyzed (Participants) | 162
Score on a scale
  Month 3: number analyzed (Participants) | 115
  Month 3 | 0.2 (15.52)
  Month 6: number analyzed (Participants) | 112
  Month 6 | 0.7 (16.58)
  Month 12: number analyzed (Participants) | 102
  Month 12 | -1.4 (18.70)
  Month 18: number analyzed (Participants) | 88
  Month 18 | -0.7 (18.45)
  Month 24: number analyzed (Participants) | 38
  Month 24 | -3.2 (22.51)

9. Secondary Outcome: Change From Baseline in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core-30 (EORTC QLQ-C30): Role Functioning
Description: The EORTC QLQ-C30 is a patient completed 30 item questionnaire that is composed of both multi-item scales and single-item measures. These include five functional scales, three symptom scales, six single items and a global health status/QoL scale.
  For the role functioning scale, participants self-rated how much they were limited in doing work or daily activities, or in pursuing hobbies or other leisure time activities during the past week. The role functioning scale had 4 possible scores (1=not at all, 2=a little, 3=quite a bit, 4=very much). Scores were averaged and transformed to 0 to 100. Higher scores indicate better functioning. A positive change from baseline indicates improvement in role functioning.
Time Frame: Baseline, month 3, month 6, month 12, month 18 and month 24
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Nilotinib
Number analyzed (Participants) | 162
Score on a scale
  Month 3: number analyzed (Participants) | 115
  Month 3 | -0.1 (33.22)
  Month 6: number analyzed (Participants) | 111
  Month 6 | 2.0 (29.19)
  Month 12: number analyzed (Participants) | 102
  Month 12 | 0.5 (32.11)
  Month 18: number analyzed (Participants) | 87
  Month 18 | 0.4 (34.57)
  Month 24: number analyzed (Participants) | 38
  Month 24 | 0.4 (35.41)

10. Secondary Outcome: Change From Baseline in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core-30 (EORTC QLQ-C30): Emotional Functioning
Description: The EORTC QLQ-C30 is a patient completed 30 item questionnaire that is composed of both multi-item scales and single-item measures. These include five functional scales, three symptom scales, six single items and a global health status/QoL scale.
  For the emotional functioning scale, participants self-rated how much they felt tense, worried, irritable or depressed during the past week. The emotional functioning scale had 4 possible scores (1=not at all, 2=a little, 3=quite a bit, 4=very much). Scores were averaged and transformed to 0 to 100. Higher scores indicate better functioning. A positive change from baseline indicates improvement in emotional functioning.
Time Frame: Baseline, month 3, month 6, month 12, month 18 and month 24
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Nilotinib
Number analyzed (Participants) | 162
Score on a scale
  Month 3: number analyzed (Participants) | 114
  Month 3 | 8.1 (20.73)
  Month 6: number analyzed (Participants) | 110
  Month 6 | 8.6 (22.06)
  Month 12: number analyzed (Participants) | 101
  Month 12 | 7.2 (25.59)
  Month 18: number analyzed (Participants) | 85
  Month 18 | 4.7 (24.48)
  Month 24: number analyzed (Participants) | 38
  Month 24 | 0.0 (21.14)

11. Secondary Outcome: Change From Baseline in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core-30 (EORTC QLQ-C30): Cognitive Functioning
Description: The EORTC QLQ-C30 is a patient completed 30 item questionnaire that is composed of both multi-item scales and single-item measures. These include five functional scales, three symptom scales, six single items and a global health status/QoL scale.
  For the cognitive functioning scale, participants self-rated the extent of difficulty in concentrating on things or remembering things during the past week. The cognitive functioning scale had 4 possible scores (1=not at all, 2=a little, 3=quite a bit, 4=very much). Scores were averaged and transformed to 0 to 100. Higher scores indicate better functioning. A positive change from baseline indicates improvement in cognitive functioning.
Time Frame: Baseline, month 3, month 6, month 12, month 18 and month 24
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Nilotinib
Number analyzed (Participants) | 162
Score on a scale
  Month 3: number analyzed (Participants) | 114
  Month 3 | -2.3 (20.67)
  Month 6: number analyzed (Participants) | 110
  Month 6 | -3.8 (23.10)
  Month 12: number analyzed (Participants) | 101
  Month 12 | -7.1 (24.65)
  Month 18: number analyzed (Participants) | 85
  Month 18 | -8.0 (27.77)
  Month 24: number analyzed (Participants) | 38
  Month 24 | -8.3 (28.67)

12. Secondary Outcome: Change From Baseline in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core-30 (EORTC QLQ-C30): Social Functioning
Description: The EORTC QLQ-C30 is a patient completed 30 item questionnaire that is composed of both multi-item scales and single-item measures. These include five functional scales, three symptom scales, six single items and a global health status/QoL scale.
  For the social functioning scale, participants self-rated how much their physical condition or medical treatment interfered with their family life and social activities during the past week. The social functioning scale had 4 possible scores (1=not at all, 2=a little, 3=quite a bit, 4=very much). Scores were averaged and transformed to 0 to 100. Higher scores indicate better functioning. A positive change from baseline indicates improvement in social functioning.
Time Frame: Baseline, month 3, month 6, month 12, month 18 and month 24
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Nilotinib
Number analyzed (Participants) | 162
Score on a scale
  Month 3: number analyzed (Participants) | 114
  Month 3 | -0.7 (26.83)
  Month 6: number analyzed (Participants) | 110
  Month 6 | 0.3 (26.03)
  Month 12: number analyzed (Participants) | 100
  Month 12 | -1.2 (27.95)
  Month 18: number analyzed (Participants) | 85
  Month 18 | -1.2 (28.15)
  Month 24: number analyzed (Participants) | 38
  Month 24 | -9.2 (28.13)

13. Secondary Outcome: Change From Baseline in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Chronic Myeloid Leukemia Specific 24 (EORTC QLQ-CML 24): Symptom Burden
Description: The EORTC QLQ-CML 24 is an internationally developed disease specific health-related quality of life questionnaire for CML patients. The questionnaire is composed of four multi-item scales and two single-item scales. The module consists of 24 items assessing symptoms burden (13 items), impact on worry/mood (4 items), impact on daily life (3 items), satisfaction with care and information (2 items) body image problems (1 item) and satisfaction with social life (1 item). The items were measured on four levels: 1=not at all, 2=a little, 3=quite a bit, 4=very much. For each domain, scores were averaged and transformed to 0 to 100. A higher score in symptom burden domain indicates a worse outcome. A negative change from baseline indicates improvement.
Time Frame: Baseline, month 3, month 6, month 12, month 18 and month 24
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Nilotinib
Number analyzed (Participants) | 162
Score on a scale
  Month 3: number analyzed (Participants) | 104
  Month 3 | 2.9 (13.90)
  Month 6: number analyzed (Participants) | 105
  Month 6 | 2.4 (13.76)
  Month 12: number analyzed (Participants) | 95
  Month 12 | 3.6 (14.29)
  Month 18: number analyzed (Participants) | 79
  Month 18 | 2.5 (12.85)
  Month 24: number analyzed (Participants) | 38
  Month 24 | 3.2 (14.46)

14. Secondary Outcome: Change From Baseline in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Chronic Myeloid Leukemia Specific 24 (EORTC QLQ-CML 24): Impact on Worry/Mood
Description: The EORTC QLQ-CML 24 is an internationally developed disease specific health-related quality of life questionnaire for CML patients. The questionnaire is composed of four multi-item scales and two single-item scales. The module consists of 24 items assessing symptoms burden (13 items), impact on worry/mood (4 items), impact on daily life (3 items), satisfaction with care and information (2 items) body image problems (1 item) and satisfaction with social life (1 item). The items were measured on four levels: 1=not at all, 2=a little, 3=quite a bit, 4=very much. For each scale, scores were averaged and transformed to 0 to 100. A higher score in impact on worry/mood domain indicates a worse outcome. A negative change from baseline indicates improvement.
Time Frame: Baseline, month 3, month 6, month 12, month 18 and month 24
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Nilotinib
Number analyzed (Participants) | 162
Score on a scale
  Month 3: number analyzed (Participants) | 104
  Month 3 | -3.4 (27.01)
  Month 6: number analyzed (Participants) | 105
  Month 6 | -4.7 (26.04)
  Month 12: number analyzed (Participants) | 95
  Month 12 | -6.0 (25.55)
  Month 18: number analyzed (Participants) | 78
  Month 18 | -3.8 (28.40)
  Month 24: number analyzed (Participants) | 38
  Month 24 | -2.0 (25.22)

15. Secondary Outcome: Change From Baseline in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Chronic Myeloid Leukemia Specific 24 (EORTC QLQ-CML 24): Impact on Daily Life
Description: The EORTC QLQ-CML 24 is an internationally developed disease specific health-related quality of life questionnaire for CML patients. The questionnaire is composed of four multi-item scales and two single-item scales. The module consists of 24 items assessing symptoms burden (13 items), impact on worry/mood (4 items), impact on daily life (3 items), satisfaction with care and information (2 items) body image problems (1 item) and satisfaction with social life (1 item). The items were measured on four levels: 1=not at all, 2=a little, 3=quite a bit, 4=very much. For each domain, scores were averaged and transformed to 0 to 100. A higher score in impact on daily life domain indicates a worse outcome. A negative change from baseline indicates improvement.
Time Frame: Baseline, month 3, month 6, month 12, month 18 and month 24
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Nilotinib
Number analyzed (Participants) | 162
Score on a scale
  Month 3: number analyzed (Participants) | 64
  Month 3 | -3.6 (25.59)
  Month 6: number analyzed (Participants) | 64
  Month 6 | -6.4 (24.07)
  Month 12: number analyzed (Participants) | 62
  Month 12 | -6.2 (26.50)
  Month 18: number analyzed (Participants) | 47
  Month 18 | -6.4 (27.87)
  Month 24: number analyzed (Participants) | 20
  Month 24 | -10.0 (31.61)

16. Secondary Outcome: Change From Baseline in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Chronic Myeloid Leukemia Specific 24 (EORTC QLQ-CML 24): Satisfaction With Care and Information
Description: The EORTC QLQ-CML 24 is an internationally developed disease specific health-related quality of life questionnaire for CML patients. The questionnaire is composed of four multi-item scales and two single-item scales. The module consists of 24 items assessing symptoms burden (13 items), impact on worry/mood (4 items), impact on daily life (3 items), satisfaction with care and information (2 items) body image problems (1 item) and satisfaction with social life (1 item). The items were measured on four levels: 1=not at all, 2=a little, 3=quite a bit, 4=very much. For each domain, scores were averaged and transformed to 0 to 100. A higher score in satisfaction with care and information domain indicates a higher level of satisfaction. A positive change from baseline indicates increasing satisfaction.
Time Frame: Baseline, month 3, month 6, month 12, month 18 and month 24
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Nilotinib
Number analyzed (Participants) | 162
Score on a scale
  Month 3: number analyzed (Participants) | 62
  Month 3 | 4.3 (30.47)
  Month 6: number analyzed (Participants) | 60
  Month 6 | 5.6 (33.71)
  Month 12: number analyzed (Participants) | 60
  Month 12 | -0.6 (34.30)
  Month 18: number analyzed (Participants) | 46
  Month 18 | 2.2 (30.35)
  Month 24: number analyzed (Participants) | 19
  Month 24 | 12.3 (30.35)

17. Secondary Outcome: Change From Baseline in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Chronic Myeloid Leukemia Specific 24 (EORTC QLQ-CML 24): Body Image Problems
Description: The EORTC QLQ-CML 24 is an internationally developed disease specific health-related quality of life questionnaire for CML patients. The questionnaire is composed of four multi-item scales and two single-item scales. The module consists of 24 items assessing symptoms burden (13 items), impact on worry/mood (4 items), impact on daily life (3 items), satisfaction with care and information (2 items) body image problems (1 item) and satisfaction with social life (1 item). The items were measured on four levels: 1=not at all, 2=a little, 3=quite a bit, 4=very much. For each domain, scores were averaged and transformed to 0 to 100. A higher score in body image problems domain indicates a worse outcome. A negative change from baseline indicates improvement.
Time Frame: Baseline, month 3, month 6, month 12, month 18 and month 24
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Nilotinib
Number analyzed (Participants) | 162
Score on a scale
  Month 3: number analyzed (Participants) | 63
  Month 3 | 2.1 (32.72)
  Month 6: number analyzed (Participants) | 64
  Month 6 | 3.1 (28.92)
  Month 12: number analyzed (Participants) | 62
  Month 12 | 7.0 (28.40)
  Month 18: number analyzed (Participants) | 47
  Month 18 | 5.7 (31.33)
  Month 24: number analyzed (Participants) | 20
  Month 24 | 3.3 (35.71)

18. Secondary Outcome: Change From Baseline in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Chronic Myeloid Leukemia Specific 24 (EORTC QLQ-CML 24): Satisfaction With Social Life
Description: The EORTC QLQ-CML 24 is an internationally developed disease specific health-related quality of life questionnaire for CML patients. The questionnaire is composed of four multi-item scales and two single-item scales. The module consists of 24 items assessing symptoms burden (13 items), impact on worry/mood (4 items), impact on daily life (3 items), satisfaction with care and information (2 items) body image problems (1 item) and satisfaction with social life (1 item). The items were measured on four levels: 1=not at all, 2=a little, 3=quite a bit, 4=very much. For each domain, scores were averaged and transformed to 0 to 100. A higher score in satisfaction with social life domain indicates a higher level of satisfaction. A positive change from baseline indicates increasing satisfaction.
Time Frame: Baseline, month 3, month 6, month 12, month 18 and month 24
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Nilotinib
Number analyzed (Participants) | 162
Score on a scale
  Month 3: number analyzed (Participants) | 60
  Month 3 | 3.9 (34.22)
  Month 6: number analyzed (Participants) | 62
  Month 6 | 9.7 (39.76)
  Month 12: number analyzed (Participants) | 61
  Month 12 | 6.6 (41.19)
  Month 18: number analyzed (Participants) | 47
  Month 18 | 8.5 (39.60)
  Month 24: number analyzed (Participants) | 19
  Month 24 | 14.0 (30.05)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from first dose of study treatment until end of study treatment plus 30 days post treatment, up to maximum duration of 25 months
Description: Any sign or symptom that occurs during the study treatment plus the 30 days post treatment. Safety analysis population included all participants who received at least one dose of study drug and had at least one post-baseline safety assessment. Of note, the statement that a patient had no adverse events also constituted a safety assessment.
Arm/Group | Nilotinib
All-Cause Mortality (participants affected / at risk) | 1/171
Serious Adverse Events (participants affected / at risk) | 38/171
Other Adverse Events (participants affected / at risk) | 148/171
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nilotinib (N=171)
Anaemia (Blood and lymphatic system disorders) | 1
Blood loss anaemia (Blood and lymphatic system disorders) | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 2
Angina pectoris (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Cardiac arrest (Cardiac disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 1
Coronary artery disease (Cardiac disorders) | 2
Coronary artery occlusion (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Sinus node dysfunction (Cardiac disorders) | 1
Tachyarrhythmia (Cardiac disorders) | 1
Visual impairment (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Gastritis (Gastrointestinal disorders) | 2
Haemorrhoids thrombosed (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 1
General physical health deterioration (General disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Pain (General disorders) | 1
COVID-19 (Infections and infestations) | 1
Infectious pleural effusion (Infections and infestations) | 1
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 1
Soft tissue infection (Infections and infestations) | 1
Craniocerebral injury (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 1
Fracture displacement (Injury, poisoning and procedural complications) | 1
Postoperative ileus (Injury, poisoning and procedural complications) | 1
Rib fracture (Injury, poisoning and procedural complications) | 1
Troponin increased (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Spinal pain (Musculoskeletal and connective tissue disorders) | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Oral papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Squamous cell carcinoma of the vulva (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Transformation to acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Facial nerve disorder (Nervous system disorders) | 1
IIIrd nerve paralysis (Nervous system disorders) | 1
Loss of consciousness (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Depression (Psychiatric disorders) | 2
Acute kidney injury (Renal and urinary disorders) | 1
Renal colic (Renal and urinary disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Ureterolithiasis (Renal and urinary disorders) | 1
Urinary incontinence (Renal and urinary disorders) | 1
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1
Extremity necrosis (Vascular disorders) | 1
Hypertension (Vascular disorders) | 1
Peripheral arterial occlusive disease (Vascular disorders) | 3
Peripheral vascular disorder (Vascular disorders) | 1
Thrombosis (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nilotinib (N=171)
Thrombocytopenia (Blood and lymphatic system disorders) | 15
Abdominal pain (Gastrointestinal disorders) | 11
Abdominal pain upper (Gastrointestinal disorders) | 17
Constipation (Gastrointestinal disorders) | 14
Diarrhoea (Gastrointestinal disorders) | 20
Dyspepsia (Gastrointestinal disorders) | 10
Nausea (Gastrointestinal disorders) | 20
Fatigue (General disorders) | 34
Oedema peripheral (General disorders) | 10
Pyrexia (General disorders) | 11
Nasopharyngitis (Infections and infestations) | 31
Alanine aminotransferase increased (Investigations) | 12
Gamma-glutamyltransferase increased (Investigations) | 9
Hypercholesterolaemia (Metabolism and nutrition disorders) | 14
Arthralgia (Musculoskeletal and connective tissue disorders) | 22
Back pain (Musculoskeletal and connective tissue disorders) | 18
Muscle spasms (Musculoskeletal and connective tissue disorders) | 15
Myalgia (Musculoskeletal and connective tissue disorders) | 11
Dizziness (Nervous system disorders) | 11
Headache (Nervous system disorders) | 29
Cough (Respiratory, thoracic and mediastinal disorders) | 10
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 13
Alopecia (Skin and subcutaneous tissue disorders) | 25
Dry skin (Skin and subcutaneous tissue disorders) | 18
Pruritus (Skin and subcutaneous tissue disorders) | 37
Rash (Skin and subcutaneous tissue disorders) | 26
Hypertension (Vascular disorders) | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial

DOCUMENTS (2):
  • Study Protocol (2021-02-15): https://cdn.clinicaltrials.gov/large-docs/74/NCT02546674/Prot_000.pdf
  • Statistical Analysis Plan (2021-11-19): https://cdn.clinicaltrials.gov/large-docs/74/NCT02546674/SAP_001.pdf